CLINICAL TRIAL: NCT03219944
Title: Clinical Evaluation of Platelet Rich Fibrin Versus Subepithelial Connective Tissue Graft for Soft Tissue Augmentation Around Implant in the Aesthetic Zone: A Randomized Control Clinical Trial
Brief Title: Clinical Evaluation of Platelet Rich Fibrin Versus Subepithelial Connective Tissue Graft for Soft Tissue Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, may mohamed kamal, master student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PERIODONTOLOGYcairo university
Record Dates: First submitted 2017-07-10; First posted 2017-07-18 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Patients With at Least Single Missing Anterior Tooth; Thin Gingival Biotype

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Fibrin for soft tissue augmentation (Experimental): blood will be drawn from the patient vein for PRF. The blood sample will be centrifuged for 10-12 min. PRF membrane is obtained
  Interventions: Procedure: Platelet Rich Fibrin
- sub epithelial connective tissue graft (Active Comparator): The connective tissue graft will be harvested from the palate. Then the SCTG will be placed over the recipient site extending palataly and sutured.
  Interventions: Procedure: sub epithelial connective tissue graft

INTERVENTIONS:
Procedure: Platelet Rich Fibrin — : Platelet Rich Fibrin for soft tissue augmentation around implant in the aesthetic zone
  Arms: Platelet Rich Fibrin for soft tissue augmentation
Procedure: sub epithelial connective tissue graft — sub epithelial connective tissue graft for soft tissue augmentation around implant in the aesthetic zone
  Arms: sub epithelial connective tissue graft

SUMMARY:
Soft tissue biotype is a critical factor for success of implant in the esthetic zone . Different soft tissue augmentation techniques have been employed to increase soft tissue thickness such as: autogenous grafts, allografts, xenografts and living cellular construct (LCC). Studies showed that, allografts and xenografts were inferior when compared with autogenous graft . However, few studies were conducted to evaluate the efficacy of soft tissue augmentation with platelet rich fibrin in order to overcome the patient morbidity with SCTG.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with missing maxillary anterior toot teeth.
2. Thin gingival biotype.
3. Adequate inter-arch space for placement of the implant prosthetic part.
4. Good oral hygiene where gingival index is (0, 1) (Loe and Silness 1963).

Exclusion Criteria:

1. Patient with medical condition that is contraindicated with the surgical procedure
2. Patients receiving treatment that affect the healing ability.
3. Patients with local pathological defects related to the area of interest.
4. Smokers or pregnant women.
5. Patients with parafunctional habits that may jeopardize the implant longevity and affect the results of the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-08-15 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Crestal bone resorption | 6 months
  measured mesially and distally using periapical xray in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Maymohamedkamal, Cairo, Elmaniel, Egypt